CLINICAL TRIAL: NCT02055339
Title: Comparison of Nasal Continuous Positive Airway Pressure With Low Flow Oxygen Versus Heated, Humidified High Flow Nasal Cannula for Oral Feeding of the Premature Infant (CHOMP Trial): A Pilot Study
Brief Title: Pilot Study Comparing Different Modes of Non-invasive Ventilation for the Oral Feeding of Preterm Infants
Acronym: CHOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Sandra Leibel, Lecturer, Neonatologist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MountSinaiH
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Feeding Behavior; Chronic Lung Disease
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fisher & Paykel heated humidified high flow nasal cannula (Experimental): For neonates randomized to HHHFNC, they will be placed on a flow rate equivalent to the pressures of nCPAP they were originally receiving based on a published chart, or stay on the same flow rate prior to randomization. When it is time for oral feeds, the Registered Nurse (RN) will turn the dial of the high flow circuit down to 2 lpm. The baby will then proceed to feed for up to one hour, and afterwards, will be turned back up to the flow rate they were on prior to feeds.
  Interventions: Device: Fisher & Paykel heated humidified high flow nasal cannula
- InfantFlow/RAM nasal continuous positive airway pressure (Active Comparator): Neonates randomized to the nCPAP arm will remain on the nCPAP pressures they were on before recruitment into the study or match the flow rate they were receiving on high flow based on a published chart. The nCPAP circuit will only be removed when it is time for oral feeds. The respiratory therapist (RT) will exchange the circuit for a low flow nasal cannula which will be set at the flow that is optimal for the baby's gestational age saturations. The baby will then proceed to feed for up to one hour, and afterwards, will be changed back to the nCPAP circuit.
  Interventions: Device: InfantFlow/RAM nasal continuous positive airway pressure

INTERVENTIONS:
Device: Fisher & Paykel heated humidified high flow nasal cannula
  Arms: Fisher & Paykel heated humidified high flow nasal cannula
Device: InfantFlow/RAM nasal continuous positive airway pressure
  Arms: InfantFlow/RAM nasal continuous positive airway pressure

SUMMARY:
Preterm infants born before 28 weeks gestation are at risk for lung disease and require oxygen and pressure to keep their lungs open. This usually involves a device called nasal continuous positive airway pressure (nCPAP). When preterm babies reach a certain age, they are ready to begin to feed by mouth, but for those on nCPAP, oral feeds are usually not started due to concerns for choking. This may cause them to miss their window of learning and may lead to a longer hospital stay or oral aversion. Sometimes babies are switched from nCPAP to low flow oxygen (LFO2) for a short time for oral feeds, but this may not provide enough support for their lungs. Heated, humidified high flow nasal cannula (HHHFNC) is another mode of providing oxygen and pressure. It is equal to nCPAP in small babies transitioning off of ventilators, but no studies have been done in older babies. We plan to compare the feeding of babies orally using either nCPAP with LFO2 or HHHFNC in preterm babies born before 28 weeks gestation who are now 34 weeks corrected gestational age. The goal will be the fastest time to full oral feeds.

DETAILED DESCRIPTION:
The primary objective of this study is to assess whether a baby born at less than 28 weeks gestation who at 34 weeks corrected gestational age, will reach full oral feeds faster on the current practice of nasal continuous positive airway pressure (nCPAP) and low flow oxygen (LFO2) or the new intervention of heated, humidified high flow nasal cannula (HHHFNC).

The specific aim of this study is to investigate the effectiveness and safety of using nCPAP and LFO2 versus HHHFNC for reaching full oral feeds in premature infants.

We hypothesize that the use of HHHFNC at the initiation of oral feeding will allow babies to reach full feeds sooner as compared with nCPAP and LFO2.

Babies born at extreme prematurity (<28 weeks gestation), are at risk of chronic lung disease due to lung immaturity. A proportion of preterm infants remains dependent on non-invasive ventilation at the corrected gestational age when they are at the neurodevelopmental stage of oral feeds. If oral feeds are not initiated in a timely manner, delays in progression of oral feeds and oral aversion may occur, resulting in longer hospital stays and/or gastrostomy tube insertions. Those that are nCPAP dependant are unable to orally feed due to safety concerns so are placed on a low pressure system of low flow nasal cannula during feeds. This may lead to microatelectasis in those babies needing a higher pressure to maintain gas exchange. HHHFNC is another method of non-invasive ventilation and it can be changed from a high pressure system (in litres per minute) to a low pressure system by turning a dial, and not having to disconnect the baby from the respiratory system.

Randomized controlled trial consisting of two arms: 1) The CPAP/LFO2 arm in which the babies will be maintained on nCPAP until the time of oral feeds wherein they will have their circuits exchanged for a low flow cannula. 2) The HHHFNC arm in which babies will be maintained on 5 lpm of HHHFNC until the time of oral feeds, wherein they will have their flows turned down to 2 lpm. The study will be conducted in a level III neonatal intensive care unit (NICU) in Mount Sinai hospital. The study subjects are 40 preterm babies that were born before 28 weeks gestational age who are now 34 weeks corrected gestational age (CGA), which are dependent on non-invasive ventilation and are receiving full feeds via nasogastric tube. The randomization will occur at 33+6/7 weeks CGA. Demographic characteristics will be compared between groups using Chi-square test or Fisher's exact test for categorical variables. Differences between continuous variables will be assessed using Student's t-test or Mann-Whitney U test for non-normally distributed variables. The primary outcome (time to full oral feeds) is a binary outcome and will be compared between groups using Chi-square test or Fisher's exact test. A difference of a p-value of <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of <28 weeks (24+0 to 27+6) with corrected gestational age of 34 weeks
* Neonates requiring respiratory support in the form of nCPAP or HHHFNC at any pressure at 34 weeks corrected gestational age and failing a trial of low flow oxygen or room air
* Full enteral feeding tolerated through a nasogastric tube

Exclusion Criteria:

* Gestational age > 28 weeks
* Neonate requiring biphasic nCPAP
* Mother never at the bedside and no consent for bottle feeds
* Severe nasal breakdown or genetic/neurologic abnormalities which impair oral feeding

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to reach full oral feeds | 2 months

SECONDARY OUTCOMES:
Time on non-invasive ventilation or oxygen | 2 months
Occurrence of feeding intolerance or reflux | 2 months
Occurrence of apneas/bradycardias/desaturations above baseline | 2 months
Weight gain | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Leibel, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital NICU, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Leibel SL, Castro M, McBride T, Hassall K, Sarmiento K, Ye XY, Shah V. Comparison of Continuous positive airway pressure versus High flow nasal cannula for Oral feeding Preterm infants (CHOmP): randomized pilot study. J Matern Fetal Neonatal Med. 2022 Mar;35(5):951-957. doi: 10.1080/14767058.2020.1735339. Epub 2020 Mar 5. PMID 32138561